CLINICAL TRIAL: NCT07399457
Title: Development of a Nature-based Physical Activity Toolkit for University Counseling Centers
Brief Title: A Nature-based Physical Activity Therapy Group for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: Frontiers Clinical & Translational Science Institute (Unknown)
Responsible Party: Principal Investigator, Emily Mailey, Associate Professor, Kansas State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-12065
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Depression and Anxiety Symptom
Keywords: anxiety; college students; physical activity; nature; group therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Received the Moving Naturally Through Challenges group therapy intervention
  Interventions: Behavioral: Moving Naturally Through Challenges group therapy

INTERVENTIONS:
Behavioral: Moving Naturally Through Challenges group therapy — The intervention included 8 weeks of group therapy. Each session was 90 minutes and incorporated 30 minutes of nature-based physical activity and 60 minutes of traditional group therapy with content focused on managing anxiety.
  Other Names: nature-based physical activity therapy group

SUMMARY:
This study examined the feasibility, acceptability, and preliminary effectiveness of a nature-based physical activity group delivered by K-State Counseling and Psychological Services (CAPS) for students experiencing depression and anxiety.

DETAILED DESCRIPTION:
For this study, our research team partnered with two CAPS therapists to develop a new therapy group called Moving Naturally Through Challenges, which focused on nature-based physical activity as a tool for managing symptoms of depression and anxiety. Prior to group implementation, the researchers and therapists collaborated to develop a detailed implementation handbook with weekly lesson plans for the eight group therapy sessions. Next, we conducted a 2-hour training workshop with all CAPS staff to familiarize them with the content and empower them to refer students to the group.

This intervention was delivered as part of group therapy services offered by CAPS. Students seeking services at CAPS whose primary presenting concerns were depression and/or anxiety were encouraged to consider joining the Moving Naturally group. Interested students attended a 30-minute pre-group screening meeting with the group facilitators to ensure it was a good fit for their needs, and then signed a consent form to formalize their enrollment in the study.

The therapy group ran during the spring semester for 8 weeks. Each session lasted 1.5 hours, and included a weekly discussion topic, applied activities for students (e.g., goal setting and planning), and 30 minutes of nature-based physical activity. Activities included walking, hiking, yoga, outdoor games, resistance training, and sport-based activities that were moderate in intensity. Each participant received a Fitbit, yoga mat, resistance band, and water bottle to bring to each session. The group facilitators received training in group fitness instruction prior to leading the group sessions.

To assess changes in mental health outcomes, all students completed the Counseling Center Assessment of Psychological Symptoms upon intake at CAPS, and again upon completion of the therapy group. In addition, students rated their enjoyment of each group therapy session using the Group Session Rating Scale. Participants were asked to wear their Fitbit 24/7 (except when charging) throughout the 8-week duration of the study, and our research team is able to access their data using the Fitabase platform. Additional data and feedback were collected from the therapists who attended the training and facilitated the group.

ELIGIBILITY:
Inclusion Criteria:

* Attends an intake session at CAPS
* Passes the pre-group screening (therapist and client agree that group is a good fit for student's needs)

Exclusion Criteria:

* Medical condition that prevents safe participation in physical activity (assessed via ACSM risk screener)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Attendance | Weekly across the 8-week intervention
  The percentage of total group therapy sessions participants attended
Group enjoyment and satisfaction | Weekly across the 8-week therapy group
  Assessed using the Group Session Rating Scale. Each of the 6 items is rated on a scale from 0-10, with higher scores indicating higher group enjoyment and satisfaction with group relationships, topics, approach, activity, skills, and overall.

SECONDARY OUTCOMES:
Depression and anxiety | Baseline and week 8
  Measured via the Counseling Center Assessment of Psychological Symptoms (CCAPS). The depression, general anxiety, and social anxiety subscales are scored on a scale from 0-100, with higher scores indicating greater depression and anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data is private health information.